CLINICAL TRIAL: NCT02087306
Title: A Phase 3, Open-Label, Multicenter Study of the Safety and Efficacy of Brincidofovir (CMX001) in the Treatment of Early Versus Late Adenovirus Infection
Brief Title: Study to Assess the Safety and Efficacy of Brincidofovir in Treatment of Early Versus Late Adenovirus Infection
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Jazz Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CMX001-304
Record Dates: First submitted 2014-03-12; First posted 2014-03-14 (Estimated); Results first posted 2021-08-13 (Actual); Last update posted 2021-08-13 (Actual); Status verified 2021-07

CONDITIONS: Adenovirus Infection
Keywords: Adenovirus Infection
MeSH Terms: conditions — Adenoviridae Infections | interventions — brincidofovir

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Brincidofovir (Experimental): Subjects who weighed <50 kg received 2 mg/kg (not to exceed 100 mg) BCV twice weekly administered orally as the appropriate volume of 10-mg/mL liquid suspension.
  Subjects who weighed ≥50 kg received 100 mg BCV twice weekly administered orally as one 100 mg tablet (or the appropriate volume of 10-mg/mL liquid suspension if unable to swallow solid medicine).
  Interventions: Drug: Brincidofovir

INTERVENTIONS:
Drug: Brincidofovir — BCV administered twice weekly, dose depending on weight.
  Other Names: BCV; CMX001

SUMMARY:
This was a Phase 3 open-label, non-randomized, multicenter study of oral brincidofovir (BCV) administered twice weekly for the treatment of adenovirus (AdV) infection detected during asymptomatic AdV viremia or during symptomatic AdV infection.

DETAILED DESCRIPTION:
This was a Phase 3 open-label, non-randomized, multicenter study of the safety, tolerability, and efficacy of oral brincidofovir (BCV) when administered twice weekly for the treatment of disseminated adenovirus (AdV) disease and for the treatment of AdV infection when treatment was initiated in subjects who were at risk of progression to disseminated disease (i.e., during the asymptomatic or localized phases of infection).

ELIGIBILITY:
Inclusion Criteria Subjects were required to meet all of the following criteria, as applicable, to be eligible to participate in this study.

1. Were male or female, aged 2 months or older.
2. Had either of the following:

   * Disseminated adenovirus (AdV) disease; or
   * An underlying immunocompromised state and were at risk of progression to disseminated AdV disease.

   [Note: Subjects with symptomatic AdV infection (i.e., localized or disseminated AdV disease) could have been screening immediately, with brincidofovir (BCV) therapy initiated after receipt of the screening virology results from the designated central virology laboratory confirming study eligibility. Subjects with asymptomatic AdV infection (i.e., had no symptoms of AdV disease) could have been consented and screened only if they had at least 1 positive or detectable AdV DNA (quantitative [q]) polymerase chain reaction (PCR) test (in any blood fluid or compartment) from the local virology laboratory, with treatment initiated only after confirmation of AdV positivity by 2 separate measurements at the designated central virology laboratory. Where the results from 2 AdV DNA (q)PCR measurements in plasma or non-plasma body fluid or compartment were needed to show that a subject was at risk of progression to disseminated AdV disease, the second measurement had to be resulted prior to the initiation of BCV therapy.]
3. Were able to ingest and absorb oral medication (in the judgement of the investigator and based on lack of significant gastrointestinal [GI] events/medical history).
4. If male of reproductive potential, were willing to use an acceptable contraceptive method(s) during sexual intercourse with a female partner of reproductive potential throughout the duration of this participation in the study and for at least 6 months after his last dose of BCV.
5. If female of reproductive potential, i.e., not premenarche, postmenopausal, surgically sterile, or had documented ovarian failure, were willing to use 2 acceptable contraceptive methods, 1 of which must have been a barrier method, during sexual intercourse with a nonsterile male partner, throughout the duration of her participation in the study and for at least 6 months after her last dose of BCV.
6. Were willing and able to understand and provide written informed consent to participate in the study. [Note: If the subject was under 18 years of age or was otherwise unable to legally give his or her informed consent to participate in the study, then written informed consent to participate had to be obtained from the parent(s) or legal guardian(s) of the subject or other legal personal representative(s), as applicable. In addition, in the case of minor subjects, the written assent of the subject to participate in the study was obtained where required by applicable institutional policy on the consenting of minor study participants.]
7. The subject and his or her caregivers (as applicable) were willing and able to participate in all required study activities for the entire duration of the study (i.e., through completion of Week 36).

Exclusion Criteria

Subjects who met any of the following criteria (as applicable) were not eligible to participate in this study:

1. If a female of reproductive potential, the subject was pregnant, planning to become pregnant during the study or within 6 months after their anticipated last BCV dose, or was nursing a child.
2. Had hypersensitivity (not including renal dysfunction or eye disorder) to cidofovir (CDV) or to BCV or its formulation excipients.
3. Had received treatment with another investigational drug within 14 days prior to Day 1 unless prior approval was received from the Chimerix medical monitor (or designee).
4. Were participating in another interventional clinical trial unless prior approval was received from the Chimerix medical monitor (or designee).
5. Had previously received an anti-AdV vaccine or a cell-based anti-AdV therapy.
6. Were receiving intravenous (IV) CDV, leflunomide, vidarabine, systemic ribavirin, or another investigational anti-AdV drug at Day 1. [Note: Subjects who were receiving treatment with IV CDV prior to enrollment had to discontinue IV CDV and wait until a minimum of 48 hours had elapsed from last IV CDV administration before initiating BCV therapy. All other drugs had to be discontinued prior to Day 1.]
7. Were receiving digoxin or ketoconazole (other than topical formulations) at Day 1 or were anticipated to need treatment with either drug during the treatment phase of the study.
8. Were infected with HIV, hepatitis B virus (HBV), and/or hepatitis C virus (HCV), had evidence of active viral replication within 6 months prior to screening, as demonstrated by detectable HIV or HCV RNA, or had detectable HBV DNA in blood, plasma or serum.
9. Had end-stage renal disease, i.e., an estimated glomerular filtration rate <15 mL/min, unless receiving renal replacement therapy.
10. Had a serum alanine aminotransferase or aspartate aminotransferase concentration >5 x the upper limit of normal (ULN), or a serum total bilirubin concentration >2 x the ULN and a serum direct (conjugated) bilirubin concentration >1.5 x the ULN, as reported by the central safety laboratory, unless, in the judgment of the investigator, the abnormality(ies) was/were related to the subject's AdV infection/disease.
11. Had ongoing Grade 3 or higher diarrhea, unless, in the judgment of the investigator, the diarrhea was related to the subject's underlying AdV infection/disease.
12. Had Stage 3 or higher graft versus host disease (GVHD) of the intestine (GI-GVHD or any other GI disease that would have, in the judgment of the investigator, precluded the subject from taking or absorbing oral medication (e.g., clinically active Crohn's disease, ischemic colitis, moderate or severe ulcerative colitis, small bowel resection, ileus, or any condition expected to require abdominal surgery during the course of study participation).
13. Had any other condition, including abnormal laboratory values, that would have, in the judgment of the investigator, put the subject at increased risk by participating in the study, or would have interfered with the conduct or planned analyses of the study.

Min Age: 2 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 201 (Actual)
Dates: Start 2014-03 (Actual); Primary Completion 2016-06 (Actual); Study Completion 2016-08 (Actual)

CONTACTS AND LOCATIONS:
Locations (33):
- United States (33):
  - Phoenix Children's Hospital, Phoenix, Arizona
  - Children's Hospital Los Angeles, Los Angeles, California
  - Stanford Children's Hospital, Palo Alto, California
  - Stanford University, Stanford, California
  - Children's Hospital Colorado, Aurora, Colorado
  - Children's National Health System, Washington D.C., District of Columbia
  - Children's Healthcare of Atlanta, Aflac Cancer and Blood Center, Atlanta, Georgia
  - Ann & Robert H. Lurie Children's Hospital of Chicago, Chicago, Illinois
  - University of Chicago, Chicago, Illinois
  - Children's Hospital, New Orleans, Louisiana
  - Johns Hopkins University, Baltimore, Maryland
  - Brigham and Woman's Hospital, Boston, Massachusetts
  - University of Minnesota, Minneapolis, Minnesota
  - Children's Mercy Hospital, Kansas City, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - University of Nebraska, Omaha, Nebraska
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Weill Cornell Medical College/ New York Presbyterian Hospital, New York, New York
  - Montifore Medical Center, The Bronx, New York
  - Levine Children's Hospital, Charlotte, North Carolina
  - Duke University Medical Center, Durham, North Carolina
  - Cincinnati Children's Hospital, Cincinnati, Ohio
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Children's Hospital of Pittsburgh, Pittsburgh, Pennsylvania
  - St. Jude Children's Hospital, Memphis, Tennessee
  - Cook Children's Medical Center, Fort Worth, Texas
  - Baylor College of Medicine, Houston, Texas
  - MD Anderson Cancer Center, Houston, Texas
  - Intermountain Healthcare Research, Salt Lake City, Utah
  - University of Utah Huntsman Cancer Institute, Salt Lake City, Utah
  - Fred Hutchingson Cancer Center, Seattle, Washington
  - Seattle Children's Hospital, Seattle, Washington
  - Medical College of Wisconsin, Milwaukee, Wisconsin

RESULTS

PARTICIPANT FLOW:
Groups:
- Cohort A: Allogeneic hematopoietic cell transplant recipients at risk of progression to disseminated adenovirus (AdV) disease (i.e., subjects with either asymptomatic AdV infection or localized adenovirus disease) and who weighed ≤120 kg.
  Subjects who weighed <50 kg received 2 mg/kg (not-to-exceed 100 mg) brincidofovir (BCV) twice weekly, administered orally as the appropriate volume of 10-mg/mL liquid suspension.
  Subjects who weighed ≥50 kg received BCV 100 mg twice weekly, administered orally as one 100-mg tablet (or the appropriate volume of 10-mg/mL liquid suspension if unable to swallow solid medicine).
- Cohort B: Allogeneic hematopoietic cell transplant recipients with disseminated adenovirus disease who weigh ≤120 kg.
  Subjects who weighed <50 kg received 2 mg/kg brincidofovir (BCV; not to exceed 100 mg) twice weekly, administered orally as the appropriate volume of 10-mg/mL liquid suspension.
  Subjects who weighed ≥50 kg received 100 mg BCV twice weekly, administered orally as one 100 mg tablet (or the appropriate volume of 10-mg/mL liquid suspension if unable to swallow solid medicine).
- Cohort C: Allogeneic hematopoietic cell transplant recipients who weighed >120 kg and all other immunocompromised subjects with disseminated adenovirus (AdV) disease or subjects who were at risk of progression to disseminated AdV disease, as well as non-immunocompromised subjects with disseminated AdV disease.
  Subjects who weighed <50 kg received 2 mg/kg (not to exceed 100 mg) brincidofovir (BCV) twice weekly, administered orally as the appropriate volume of 10-mg/mL liquid suspension.
  Subjects who weighed ≥50 kg received 100 mg BCV twice weekly, administered orally as one 100-mg tablet (or the appropriate volume of 10-mg/mL liquid suspension if unable to swallow solid medicine).
Period: Overall Study
Arm/Group | Cohort A | Cohort B | Cohort C
Started | 65 | 93 | 43
Completed | 29 | 29 | 16
Not Completed | 36 | 64 | 27

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cohort A | Cohort B | Cohort C | Total
Number analyzed (Participants) | 65 | 93 | 43 | 201
Age, Continuous [Mean (Standard Deviation); unit: years] | 19 (17.4) | 20 (23.1) | 17 (21.9) | 19 (21.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 26 | 30 | 16 | 72
  Male | 39 | 63 | 27 | 129

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With All-Cause Mortality
Description: The primary efficacy endpoint was the evaluation of the effect of brincidofovir (BCV) on all-cause mortality when used for the treatment of disseminated adenovirus (AdV) disease in all hematopoietic cell transplant (HCT) recipients. The primary endpoint associated with this objective was all-cause mortality through Day 60.
Time Frame: 60 days
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort A | Cohort B | Cohort C
Number analyzed (Participants) | 65 | 93 | 43
Participants | 9 | 27 | 8

2. Secondary Outcome: Number of Participants With Reduction in Adenovirus Viremia
Description: A secondary endpoint was the evaluation of virologic response (plasma adenovirus [AdV] DNA viremia) to brincidofovir treatment. Blood (plasma) was collected at screening, before dosing on Day 1 (to establish baseline), and at each subsequent assessment during the treatment and post-treatment phases for the analysis of AdV DNA viremia. All samples collected for analysis of AdV were analyzed by the designated central virology laboratory using proprietary real-time quantitative polymerase chain reaction (qPCR) assays. AdV in plasma were analyzed using the 7500 AdV qPCR Test, where the standardized assay plasma ranged from 190 copies/mL to 1 X 10^10 copies/mL. A "positive or detectable" result referred to the measurement of AdV DNA at concentrations ≥190 copies/mL, a result below the lower limit of detection (LLOQ) (i.e., not detected) was imputed as 1 copy/mL, and a result below the lower limit of quantitation but detected will be imputed at 1 unit less than LLOQ (e.g., 189 copies/mL).
Time Frame: Assessed 13 weeks (through 7 days post-last BCV dose); during treatment up to 12 weeks reported
Population: Subjects with AdV viremia at baseline in the Intention-to-Treat Analysis Set. The Intention-to-Treat Analysis Set included all subjects who received at least 1 dose of BCV.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort A | Cohort B | Cohort C
Number analyzed (Participants) | 41 | 86 | 30
Participants
  Undetectable AdV viremia at any time on-treatment | 30 | 52 | 17
  Undetectable AdV viremia at last on-treatment value | 25 | 41 | 16

3. Secondary Outcome: Mean Minimum On-treatment Value log10 Copies/mL Change From Baseline
Description: as for outcome 2
Time Frame: Baseline to 12 weeks
Population: Subjects who had adenovirus viremia at baseline.
Measure: Mean (Standard Deviation); unit: log10 copies/mL
Arm/Group | Cohort A | Cohort B | Cohort C
Number analyzed (Participants) | 41 | 86 | 29
log10 copies/mL
  Minimum on-treatment value log10 copies/mL change from baseline | -2.67 (1.559) | -3.27 (2.163) | -3.11 (2.127)
  Last on-treatment value log10 copies/mL change from baseline | -2.06 (1.898) | -2.61 (2.338) | -2.87 (2.291)

ADVERSE EVENTS:
Time Frame: Adverse events that started on or after the first dose of BCV up to 7 days after the last dose of BCV (through 13 weeks) are reported.
Description: As specified in the Statistical Analysis Plan, adverse events were reported by age group (i.e., pediatric and adult) rather than by cohort to provide a more useful safety assessment. Differentiating pediatric from adult safety in this broad population was more useful than differentiating safety by cohort in this uncontrolled setting.
Groups:
- Pediatric: Subjects aged 2 months to <18 years.
- Adult: Subjects aged ≥18 years
Arm/Group | Pediatric | Adult
Serious Adverse Events (participants affected / at risk) | 93/130 | 58/71
Other Adverse Events (participants affected / at risk) | 127/130 | 71/71
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Pediatric (N=130) | Adult (N=71)
Septic shock (Infections and infestations) | 8 | 23
Adenovirus infection (Infections and infestations) | 3 | 5
Staphylococcal bacteraemia (Infections and infestations) | 6 | 0
BK virus infection (Infections and infestations) | 2 | 3
Device-related infection (Infections and infestations) | 4 | 1
Pneumonia (Infections and infestations) | 2 | 2
Sepsis (Infections and infestations) | 1 | 3
Clostridium difficile colitis (Infections and infestations) | 2 | 1
Escherichia baceraemia (Infections and infestations) | 1 | 2
Klebsiella sepsis (Infections and infestations) | 3 | 0
Rhinovirus infection (Infections and infestations) | 3 | 0
Staphylococcal infection (Infections and infestations) | 3 | 0
Candida infection (Infections and infestations) | 1 | 1
Cystitis viral (Infections and infestations) | 1 | 1
Cytomegalovirus viraemia (Infections and infestations) | 0 | 2
Enterococcal bacteraemia (Infections and infestations) | 2 | 0
Enterovirus infection (Infections and infestations) | 2 | 0
Fungal infection (Infections and infestations) | 2 | 0
Klebsiella bacteraemia (Infections and infestations) | 2 | 0
Klebsiella infection (Infections and infestations) | 2 | 0
Otitis media acute (Infections and infestations) | 1 | 1
Pneumonia adenoviral (Infections and infestations) | 0 | 2
Pseudomonas infection (Infections and infestations) | 1 | 1
Viral haemorrhagic cystitis (Infections and infestations) | 0 | 2
Zygomycosis (Infections and infestations) | 2 | 0
Acinetobacter infection (Infections and infestations) | 1 | 0
Acute sinusitis (Infections and infestations) | 1 | 0
Adenoviral hepatitis (Infections and infestations) | 1 | 0
Bacillus bacteraemia (Infections and infestations) | 1 | 0
Bacterial infection (Infections and infestations) | 1 | 0
Bronchopulmonary aspergillosis (Infections and infestations) | 1 | 0
Candida pneumonia (Infections and infestations) | 1 | 0
Candida sepsis (Infections and infestations) | 1 | 0
Cerebral toxoplasmosis (Infections and infestations) | 0 | 1
Clostridium bacteraemia (Infections and infestations) | 1 | 0
Clostridium difficile infection (Infections and infestations) | 0 | 1
Cronobacter infection (Infections and infestations) | 1 | 0
Cystitis klebsiella (Infections and infestations) | 0 | 1
Cytomegalovirus infection (Infections and infestations) | 0 | 1
Enteroabacter bacteraemia (Infections and infestations) | 1 | 0
Enterobacter sepsis (Infections and infestations) | 1 | 0
Epstein-Barr viraemia (Infections and infestations) | 1 | 0
Escherichia urinary tract infection (Infections and infestations) | 0 | 1
Eye infection bacterial (Infections and infestations) | 1 | 0
Fusarium infection (Infections and infestations) | 1 | 0
Gastroenteritis rotavirus (Infections and infestations) | 1 | 0
Listeriosis (Infections and infestations) | 1 | 0
Mastoiditis (Infections and infestations) | 0 | 1
Mycobacterium avium complex infection (Infections and infestations) | 0 | 1
Oral infection (Infections and infestations) | 1 | 0
Pancreatitis bacterial (Infections and infestations) | 1 | 0
Peritonitis (Infections and infestations) | 1 | 0
Pneumonia staphylococcal (Infections and infestations) | 1 | 0
Pneumonia streptococcal (Infections and infestations) | 0 | 1
Pseudomonal bacteraemia (Infections and infestations) | 1 | 0
Respiratory syncytial virus infection (Infections and infestations) | 1 | 0
Rotavirus infection (Infections and infestations) | 1 | 0
Soft tissue infection (Infections and infestations) | 1 | 0
Staphylococcal sepsis (Infections and infestations) | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 1 | 0
Urinary tract infection (Infections and infestations) | 1 | 0
Urinary tract infection enterococcal (Infections and infestations) | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 12 | 9
Vomiting (Gastrointestinal disorders) | 4 | 6
Abdominal pain (Gastrointestinal disorders) | 5 | 1
Nausea (Gastrointestinal disorders) | 0 | 5
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 4 | 0
Ileus (Gastrointestinal disorders) | 1 | 1
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 1
Pneumatosis intestinalis (Gastrointestinal disorders) | 2 | 0
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 2 | 0
Abdominal distension (Gastrointestinal disorders) | 1 | 0
Colitis (Gastrointestinal disorders) | 1 | 0
Duodenal ulcer perforation (Gastrointestinal disorders) | 0 | 1
Faecal volume increased (Gastrointestinal disorders) | 0 | 1
Ileal ulcer (Gastrointestinal disorders) | 1 | 0
Ileus paralytic (Gastrointestinal disorders) | 0 | 1
Pancreatitis acute (Gastrointestinal disorders) | 1 | 0
Rectal haemorrhage (Gastrointestinal disorders) | 1 | 0
Small intestinal obstruction (Gastrointestinal disorders) | 1 | 0
Acute graft versus host disease (Immune system disorders) | 25 | 14
Chronic graft versus host disease (Immune system disorders) | 0 | 4
Engraftment syndrome (Immune system disorders) | 1 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 14 | 5
Pulmonary haemorrhage (Respiratory, thoracic and mediastinal disorders) | 6 | 0
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 3 | 2
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 3 | 2
Pneumomediastinum (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Aspiration (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Diffuse alveolar damage (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Organising pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Respiratory acidosis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Respiratory depression (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Respiratory disorder (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pyrexia (General disorders) | 15 | 4
Multi-organ failure (General disorders) | 12 | 5
Asthenia (General disorders) | 0 | 1
Chest pain (General disorders) | 0 | 1
Medical device complication (General disorders) | 1 | 0
Systemic inflammatory response syndrome (General disorders) | 1 | 0
Acute kidney injury (Renal and urinary disorders) | 12 | 4
Renal failure (Renal and urinary disorders) | 3 | 2
Renal impairment (Renal and urinary disorders) | 0 | 2
Chronic kidney disease (Renal and urinary disorders) | 1 | 0
Oliguria (Renal and urinary disorders) | 1 | 0
Renal tubular acidosis (Renal and urinary disorders) | 0 | 1
Renal tubular necrosis (Renal and urinary disorders) | 0 | 1
Hypotension (Vascular disorders) | 4 | 3
Hypertension (Vascular disorders) | 1 | 3
Deep vein thrombosis (Vascular disorders) | 1 | 1
Microangiopathy (Vascular disorders) | 1 | 0
Orthostatic hypotension (Vascular disorders) | 0 | 1
Shock haemorrhagic (Vascular disorders) | 1 | 0
Visceral arterial ischaemia (Vascular disorders) | 0 | 1
Febrile neutropenia (Blood and lymphatic system disorders) | 3 | 1
Neutropenia (Blood and lymphatic system disorders) | 1 | 2
Pancytopenia (Blood and lymphatic system disorders) | 1 | 1
Thrombotic microangiopathy (Blood and lymphatic system disorders) | 1 | 1
Coagulopathy (Blood and lymphatic system disorders) | 1 | 0
Histiocytosis haematophagic (Blood and lymphatic system disorders) | 1 | 0
Lymphopenia (Blood and lymphatic system disorders) | 0 | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 1
Posterior reversible encephalopathy syndrome (Nervous system disorders) | 2 | 2
Brain mass (Nervous system disorders) | 0 | 1
Central nervous system lesion (Nervous system disorders) | 1 | 0
Cerebral ventricle dilatation (Nervous system disorders) | 1 | 0
Haemorrhagic stroke (Nervous system disorders) | 1 | 0
Metabolic encephalopathy (Nervous system disorders) | 0 | 1
Seizure (Nervous system disorders) | 1 | 0
Serotonin syndrome (Nervous system disorders) | 0 | 1
Syncope (Nervous system disorders) | 0 | 1
Wernicke's encephalopathy (Nervous system disorders) | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 3 | 2
Lactic acidosis (Metabolism and nutrition disorders) | 1 | 1
Metabolic acidosis (Metabolism and nutrition disorders) | 2 | 0
Acidosis (Metabolism and nutrition disorders) | 1 | 0
Diabetes mellitus (Metabolism and nutrition disorders) | 1 | 0
Fluid overload (Metabolism and nutrition disorders) | 1 | 0
Blood bilirubin increased (Investigations) | 6 | 0
Alanine aminotransferase increased (Investigations) | 2 | 0
Transaminases increased (Investigations) | 1 | 1
Blood potassium decreased (Investigations) | 1 | 0
Respiratory syncytial virus test positive (Investigations) | 0 | 1
Arrhythmia (Cardiac disorders) | 0 | 1
Atrial flutter (Cardiac disorders) | 0 | 1
Atrioventricular block complete (Cardiac disorders) | 1 | 0
Cardiac arrest (Cardiac disorders) | 0 | 1
Cardiac failure (Cardiac disorders) | 0 | 1
Cardio-respiratory arrest (Cardiac disorders) | 1 | 0
Left ventricular dysfunction (Cardiac disorders) | 1 | 0
Pericardial effusion (Cardiac disorders) | 1 | 0
Pericarditis (Cardiac disorders) | 0 | 1
Supraventricular tachycardia (Cardiac disorders) | 0 | 1
Tachyarrhythmia (Cardiac disorders) | 0 | 1
Tachycardia (Cardiac disorders) | 1 | 0
Acute hepatic failure (Hepatobiliary disorders) | 2 | 0
Venoocclusive liver disease (Hepatobiliary disorders) | 1 | 1
Autoimmune hepatitis (Hepatobiliary disorders) | 1 | 0
Cholelithiasis (Hepatobiliary disorders) | 1 | 0
Hepatic function abnormal (Hepatobiliary disorders) | 0 | 1
Hyperbilirubinaemia (Hepatobiliary disorders) | 1 | 0
Transplant failure (Injury, poisoning and procedural complications) | 3 | 1
Feeding tube complication (Injury, poisoning and procedural complications) | 1 | 0
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 0 | 1
Stoma complication (Injury, poisoning and procedural complications) | 1 | 0
Acute myeloid leukaemia recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 2
Leukaemia recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Post transplant lymphoproliferative disorder (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Mental status changes (Psychiatric disorders) | 1 | 2
Cataract (Eye disorders) | 1 | 0
Uveitis (Eye disorders) | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0
Myositis (Musculoskeletal and connective tissue disorders) | 1 | 0
Synovitis (Musculoskeletal and connective tissue disorders) | 1 | 0
Metachromatic leukodystrophy (Congenital, familial and genetic disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Pediatric (N=130) | Adult (N=71)
Diarrhoea (Gastrointestinal disorders) | 58 | 26
Vomiting (Gastrointestinal disorders) | 27 | 20
Abdominal pain (Gastrointestinal disorders) | 20 | 23
Nausea (Gastrointestinal disorders) | 10 | 18
Abdominal distension (Gastrointestinal disorders) | 8 | 11
Constipation (Gastrointestinal disorders) | 13 | 5
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 9 | 3
Abdominal pain upper (Gastrointestinal disorders) | 3 | 4
Colitis (Gastrointestinal disorders) | 7 | 0
Dyspepsia (Gastrointestinal disorders) | 3 | 4
Candida infection (Infections and infestations) | 8 | 7
BK virus infection (Infections and infestations) | 8 | 6
Clostridium difficile colitis (Infections and infestations) | 9 | 3
Staphylococcal bacteraemia (Infections and infestations) | 11 | 1
Pneumonia (Infections and infestations) | 5 | 6
Rhinovirus infection (Infections and infestations) | 10 | 1
Septic shock (Infections and infestations) | 8 | 3
Adenovirus infection (Infections and infestations) | 3 | 5
Alanine aminotransferase increased (Investigations) | 25 | 8
Aspartate aminotransferase increased (Investigations) | 23 | 8
Blood bilirubin increased (Investigations) | 23 | 5
Blood potassium decreased (Investigations) | 20 | 6
Blood glucose increased (Investigations) | 14 | 8
Blood magnesium decreased (Investigations) | 19 | 2
Transaminases increased (Investigations) | 8 | 6
Blood albumin decreased (Investigations) | 11 | 1
Blood sodium increased (Investigations) | 9 | 3
Blood sodium decreased (Investigations) | 9 | 2
Blood calcium decreased (Investigations) | 10 | 0
Blood potassium increased (Investigations) | 7 | 3
Gamma-glutamyltranferase increased (Investigations) | 7 | 2
Weight decreased (Investigations) | 5 | 4
Blood alkaline phosphatase increased (Investigations) | 2 | 5
Pyrexia (General disorders) | 48 | 16
Fatigue (General disorders) | 5 | 14
Multi-organ failure (General disorders) | 12 | 5
Oedema peripheral (General disorders) | 5 | 8
Asthenia (General disorders) | 1 | 4
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 17 | 5
Cough (Respiratory, thoracic and mediastinal disorders) | 9 | 8
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 8 | 7
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 5 | 9
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 6 | 7
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 7 | 4
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 7 | 3
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 7 | 1
Pulmonary haemorrhage (Respiratory, thoracic and mediastinal disorders) | 8 | 0
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 7 | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 4
Acute graft versus host disease (Immune system disorders) | 43 | 23
Chronic graft versus host disease (Immune system disorders) | 4 | 5
Decreased appetite (Metabolism and nutrition disorders) | 10 | 11
Dehydration (Metabolism and nutrition disorders) | 13 | 5
Fluid overload (Metabolism and nutrition disorders) | 10 | 3
Acute kidney injury (Renal and urinary disorders) | 22 | 7
Hypotension (Vascular disorders) | 17 | 14
Hypertension (Vascular disorders) | 12 | 7
Deep vein thrombosis (Vascular disorders) | 2 | 5
Neutropenia (Blood and lymphatic system disorders) | 16 | 7
Anaemia (Blood and lymphatic system disorders) | 7 | 2
Thrombocytopenia (Blood and lymphatic system disorders) | 4 | 4
Pancytopenia (Blood and lymphatic system disorders) | 1 | 4
Pruritus (Skin and subcutaneous tissue disorders) | 11 | 0
Rash (Skin and subcutaneous tissue disorders) | 7 | 4
Dry skin (Skin and subcutaneous tissue disorders) | 5 | 4
Depression (Psychiatric disorders) | 7 | 4
Insomnia (Psychiatric disorders) | 9 | 2
Mental status changes (Psychiatric disorders) | 3 | 6
Agitation (Psychiatric disorders) | 4 | 4
Headache (Nervous system disorders) | 4 | 4
Dizziness (Nervous system disorders) | 1 | 5
Tachycardia (Cardiac disorders) | 16 | 4
Arthralgia (Musculoskeletal and connective tissue disorders) | 9 | 3
Vision blurred (Eye disorders) | 1 | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Within 12 months after the end of the Study at all sites, if no publication of the overall multi-center results has been made, institutions are entitled to publish their locally obtained results, provided the Sponsor is given opportunity to review and comment. Institution publications may be delayed up to an additional 60 days to allow Sponsor to seek patent protection.